CLINICAL TRIAL: NCT04606134
Title: A Single Center, Prospective, Blinded Study to Evaluate the Efficacy and Safety of a Tripeptide/Hexapeptide Topical When Used With Er:YAG Hybrid Laser for the Treatment of Acne Scars
Brief Title: Tripeptide/Hexapeptide Topical and Hybrid Laser Treatment for Acne Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Mara Weinstein Velez, MD, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00003126
Record Dates: First submitted 2020-10-21; First posted 2020-10-28 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Device: Hybrid fractional laser; Other: Alastin Regenerating Skin Nectar with TriHex Technology
- Control (Placebo Comparator)
  Interventions: Device: Hybrid fractional laser; Other: Cetaphil face cream

INTERVENTIONS:
Device: Hybrid fractional laser — two treatments given one month apart
Other: Alastin Regenerating Skin Nectar with TriHex Technology — applied twice daily
  Arms: Experimental
Other: Cetaphil face cream — applied twice daily
  Arms: Control

SUMMARY:
To evaluate the efficacy of a tripeptide/hexapeptide topical (Alastin Regenerating Skin Nectar with TriHex Technology®) in wound healing and scar reduction following Erbium:YAG hybrid resurfacing laser for acne scarring compared to the standard of post-procedure care consisting of a bland moisturizer.

ELIGIBILITY:
Inclusion Criteria:

* male or females
* age 18 and older
* with evidence of grade II-III acne scars on the face (mild to moderate) as determined by the Goodman & Baron qualitative global acne scar grading system

Exclusion Criteria:

* treatment to face with any energy device within 6 months
* tanning within 7 days
* dermabrasion or chemical peel within 3 months
* current use of systemic retinoids
* keloidal scaring in the treatment area
* use of systemic steroids within 6 months
* use of topical products with retinoid, alpha-hydroxyacid, salicylic acid, vitamin C or E within 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Alastin Regenerating Skin Nectar With TriHex Technology: Hybrid fractional laser: two treatments given one month apart
  Alastin Regenerating Skin Nectar with TriHex Technology: applied twice daily
- Control: Cetaphil: Hybrid fractional laser: two treatments given one month apart
  Cetaphil face cream: applied twice daily
Period: Overall Study
Arm/Group | Experimental: Alastin Regenerating Skin Nectar With TriHex Technology | Control: Cetaphil
Started | 6 | 4
Completed | 6 | 3
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Alastin Regenerating Skin Nectar With TriHex Technology | Control: Cetaphil | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34.6 [19 to 45] | 31.5 [19 to 45] | 33.4 [19 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 3 | 7
  Asian | 1 | 1 | 2
  African American | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Erythema
Description: A colorimeter will be used to measure the erythema index. The range of the index is 0-99 with 0 indicating better outcome. Erythema will be measured at baseline and at follow-up visits. The mean change from baseline will be averaged to get the overall mean for each arm at each follow up visit.
Time Frame: baseline to day 34
Population: One participant in the control group, discontinued prior to Day 30.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 6 | 3
units on a scale | -1.687 (4.461) | 5.730 (4.461)

2. Secondary Outcome: Mean Change in Skin Barrier Function
Description: Barrier function will be measured by transepidermal water loss in grams/m2(hour). The lower the water loss the better the barrier function of the skin. Barrier function will be measured at baseline, days of laser treatment and 4 days after treatment. Laser treatment will occur at baseline and day 30. The mean change from baseline, at each follow-up visit, will be averaged to get the overall mean for each arm.
Time Frame: baseline to day 34
Population: One participant in the control group discontinued prior to second laser treatment, Day 30.
Measure: Mean (Standard Error); unit: g/m^2h
Arm/Group | Experimental | Control
Number analyzed (Participants) | 6 | 4
g/m^2h
  Day 4 | 6.502 (6.650) | 21.59 (6.650)
  Day 34: number analyzed (Participants) | 6 | 3
  Day 34 | 2.858 (7.233) | 39.07 (7.233)

3. Secondary Outcome: Number of Participants Who Scored Skin Appearance as no Change, Improved or Much Improved Using the Global Aesthetic Improvement Scale
Description: The Global Aesthetic Improvement Scale measures the appearance of the skin as reported by the participant. 1=worse; appearance has worsened compared with the original condition, 2=no change; appearance remains the same as the original condition, 3=improved; better than the initial condition, 4=much improved; marked improvement but not completely optimal, 5=very much improved; excellent or exceptional improvement. The number of participants within each grade will be reported.
Time Frame: baseline to day 90
Population: One participant in the control discontinued prior to Day 90.
Measure: Number; unit: participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 6 | 3
participants
  Improved | 4 | 1
  No Change | 2 | 1
  Much Improved | 0 | 1

4. Primary Outcome: Mean Change From Baseline in Erythema
Description: as for outcome 1
Time Frame: baseline to day 4
Population: One participant in the control group, discontinued prior to Day 30.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 6 | 4
units on a scale | 1.768 (4.218) | 5.596 (4.218)

ADVERSE EVENTS:
Time Frame: through study completion, approximately 90 days
Description: Adverse event collection did not differ from the clinicaltrials.gov definition.
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=6) | Control (N=4)
Melasma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Melasma, flare after first treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT04606134/Prot_SAP_000.pdf